CLINICAL TRIAL: NCT01183338
Title: SpO2 Accuracy Validation of Sotera Wireless Pulse Oximetry Systems During Non-Motion and Motion Conditions of Induced Hypoxia as Compared to Arterial Blood CO-Oximetry
Brief Title: Accuracy of Continuous SpO2 Measurement in Adults
Acronym: SPO2
Status: Withdrawn | Type: Observational
Sponsor: Sotera Wireless, Inc. (Industry)
Responsible Party: Gary Manning, Vice President Clinical Affairs and Business Development, Sotera Wireless, Inc.
Other Study IDs: SWI-US11-006
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: SpO2; Oxygen saturation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the accuracy of the Sotera ViSi, an investigational device, to standard devices in estimating the level of blood oxygen (SpO2) in adult human subjects.

DETAILED DESCRIPTION:
This study is a single-center blinded study that will enroll up to 15 adult subjects, male or female, of any ethnic background.

SpO2 and pulse rate measurements reported by ViSi will be compared with simultaneous measurements of blood SaO2 and pulse rate made by an FDA-cleared CO-oximeter and pulse oximeter, respectively. The paired measurements will be made in a well-controlled environment under optimal laboratory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject is a healthy volunteer capable of undergoing controlled hypoxemia to the level of 70% SaO2 (±3%) with no or minimal medical risk.
* Subject is willing and able to participate in the measurement period for up to two hours.

Exclusion Criteria:

* Subject has a carboxyhemoglobin level (COHb) ≥3%.
* Subject has a MetHb level ≥2%.
* Subject has a ctHb value ≤10g/dl.
* Subject is in another clinical study that may interfere with the results of this study.
* Subject is unable or unwilling to have a blood gas and oxygen saturation measurements taken from either wrist/hand.
* Subject is deemed by the Investigator to be medically unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers, male or female, of any ethnic background. To the extent possible while still achieving timely enrollment, subjects should vary from one another in their physical characteristics. Each subject must also meet all of the inclusion and exclusion criteria prior to study entry and give informed consent to participate in this study.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philip S. Clifford, PhD, Principal Investigator — VA Medical Center
Locations (1):
- Clinimark Desaturation Laboratory, Louisville, Colorado, United States